CLINICAL TRIAL: NCT01403922
Title: A Phase I Randomised, Placebo-Controlled, Double-Blind Study in Hypertensive Patients of the Blood Pressure Interaction Between TC-5214 and Anti-Hypertensive Medications (Calcium Channel Blockers, Beta Blockers, and ACE Inhibitors)
Brief Title: To Determine Blood Pressure Interaction Between TC-5214 and Anti-Hypertensive Medications (Calcium Channel Blockers, Beta Blockers, and ACE Inhibitors) in Patients With Chronic Hypertension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision to terminate
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D4130C00010
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Hypertension
Keywords: Phase I, Randomised, Placebo-Controlled, Double-Blind,Hypertensive Patients, Blood Pressure, Calcium Channel Blockers, Beta Blockers, ACE Inhibitors; Scientific terminology: To determine if treatment with TC5214 alone or in combination with Anti-Hypertensive Medications has an effect on sitting blood pressure; Laymen terminology: Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): TC-5214
  Interventions: Drug: TC-5214
- 2 (Experimental): TC-5214 with placebo
  Interventions: Drug: TC-5214
- 3 (Experimental): TC-5214 with placebo
  Interventions: Drug: TC-5214
- 4 (Experimental): TC-5214
  Interventions: Drug: TC-5214

INTERVENTIONS:
Drug: TC-5214 — Tablet oral bid days 1 to 7
  Arms: 1; 3
Drug: TC-5214 — Tablet oral bid days 8 to 14
  Arms: 2; 4

SUMMARY:
This is a two part study. Part 1 will determine determine if administration of TC-5214 has an effect on sitting blood pressure in patients with chronic hypertension.

Part 2 will determine any possible interactions between TC-5214 and Anti-Hypertensive Medications (Calcium Channel Blockers, Beta Blockers, and ACE Inhibitors).

DETAILED DESCRIPTION:
A Phase I Randomised, Placebo-Controlled, Double-Blind Study in Hypertensive Patients of the Blood Pressure Interaction between TC-5214 and Anti-Hypertensive Medications (Calcium Channel Blockers, Beta Blockers, and ACE Inhibitors)

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Male or female patients with chronic, stable hypertension treated for at least 1 month before screening with a calcium channel blocker, a beta blocker, or an ACE inhibitor, either as the only anti-hypertensive medication or concurrently with a diuretic. The patients should have no change in their current anti hypertensive treatment for at least 1 month before dosing
* Patients in Part 1 should have an SBP of ≤140 mmHg at screening and ≤160 mmHg at Visit 1a and pre-dose on Day 1
* Patients in Part 2 should have an SBP of ≤160 mmHg at screening Visit 1 and pre dose on Day 1. Systolic blood pressure and DBP should not vary by more than 8 mmHg and 5 mmHg, respectively, in the pre-dose period (screening, Visit 1a, and pre-dose on Day 1)
* Age 18 to 65 years (inclusive)

Exclusion Criteria:

* Other than having chronic hypertension, the history of any clinically significant medical, neurologic, or psychiatric disease or disorder which, in the opinion of the Investigator and/or the Sponsor, may either put the patient at risk because of participation in the study or influence the results, or the patient's ability to participate in the study. Patients with dyslipidaemia (diet controlled or treated with a statin) and/or metabolic syndrome (diet controlled or treated with metformin) may be entered into the study
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the investigational product
* Patients with a pre-treatment SBP (if known) of >180 mmHg or a history of accelerated or malignant hypertension based on grade III (hypertensive haemorrhages and/or cotton wool spots) or grade IV (hypertensive papilloedema) retinopathy at any time
* History or presence of gastrointestinal (including irritable bowel disease), hepatic, or renal disease (creatinine clearance of ≤50 mL/minute calculated using the Cockcroft Gault equation) or any other condition known to interfere with the ADME of the investigational product.
* Patients with a history of surgery on the gastrointestinal tract (not including appendectomy or cholecystectomy) should also be excluded
* Any significant ECG abnormality including QTcF prolongation (>450 ms) or significant arrhythmias, or junctional rhythms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Part 1: To measure the effect of TC-5214 on sitting blood pressure in patients with chronic hypertension. | Day 1 through to follow up
  The following assessments will be measured and reported:
  - A change from baseline in blood pressure and pulse rate.
Part 2: To measure the effect of TC-5214 combined with treatment with the common classes of anti-hypertensive medication (calcium channel blockers, beta blockers, angiotensin converting enzyme inhibitors) on sitting blood pressure. | Day 1 through to follow up
  The following assessments will be measured and reported:
  A change from baseline in blood pressure and pulse rate.

SECONDARY OUTCOMES:
To examine the safety and tolerability of TC-5214. | Day 1 through to Follow up
  The following assessments will be measured and reported:
  * The number of particpants with adverse events
  * A change from baseline in blood pressure and pulse rate
  * A change from baseline in laboratory assessments
  * A change from baseline in vital signs
  * A change from baseline in electrocardiogram (ECG)
  * A change from baseline in physical examination
The concentration of TC-5214 in plasma will be measured. | Day 1 to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Eriksson, MD, PhD, MBA, Study Director — AstraZeneca PharmaceuticalsKvarnbergagatan 12, 15185, Sodertalje, Sweden; James Ritter, MD,FRCP FFPM, Principal Investigator — Quintiles Drug Research Unit at Guy's HospitalQuintiles Limited6 Newcomen StreetLondon SE1 1YR
Locations (4):
- United States (2):
  - Research Site, Overland Park, Kansas
  - Research Site, Willingboro, New Jersey
- Research Site, Berlin, Germany
- Research Site, London, United Kingdom